CLINICAL TRIAL: NCT06624748
Title: Evaluation of the Opinions of Companions Who Support the Pregnant Woman During the Birth Process: Mixed Method Study
Brief Title: Companions Who Support the Pregnant Woman During the Birth Process
Acronym: SupportBirth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Bihter Akın, Assos. Prof., Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2023/1021
Record Dates: First submitted 2024-02-09; First posted 2024-10-03 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Childbirth Problems; Support, Family
Keywords: Pregnancy; Midwife

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- emotional and physical support to the pregnant woman provided by attendant (Experimental): Following the information, the attendant will provide emotional and physical support to the pregnant woman (such as massage, supporting the pregnant woman while moving, giving the pregnant woman a warm shower), and all interventions made by the companion and their duration will be recorded by the researcher in the 'Birth Process Support Form'. When the cervical dilatation is 8 cm, the Birth Comfort Scale will be applied to the pregnant woman, and two hours after the birth, the Birth Satisfaction Scale and the Postpartum Comfort Scale will be applied. Information about the birth process will be recorded in the Birth Information Form. In addition, semi-structured questions in the 'Companion Interview Form' will be asked to the companions selected for qualitative interviews and voice recording will be recorded.
  Interventions: Behavioral: emotional and physical support to the pregnant woman provided by attendant
- Standard of care (No Intervention): Women who are informed about the purpose and practices of the research and who agree to participate in the study voluntarily will not be deviated from routine practices in the hospital. Women who are followed and delivered by the same midwife will be included in the study to ensure that there is no difference between the groups in terms of episiotomy application and birth techniques. When the cervical dilatation is 8 cm, the Birth Comfort Scale will be applied to the pregnant woman, and two hours after the birth, the Birth Satisfaction Scale and the Postpartum Comfort Scale will be applied. Information about the birth process will be recorded in the Birth Information Form.

INTERVENTIONS:
Behavioral: emotional and physical support to the pregnant woman provided by attendant — The companion will provide emotional and physical support to the pregnant woman (such as massage, supporting the pregnant woman while moving, taking a warm shower, etc.), and all interventions made by the companion and their duration will be recorded by the researcher in the 'Birth Process Support Form'. When the cervical dilatation is 8 cm, the Birth Comfort Scale will be applied to the pregnant woman, and two hours after the birth, the Birth Satisfaction Scale and the Postpartum Comfort Scale will be applied. Information about the birth process will be recorded in the Birth Information Form. In addition, semi-structured questions in the 'Companion Interview Form' will be asked to the companions selected for qualitative interviews and voice recording will be recorded.
  Arms: emotional and physical support to the pregnant woman provided by attendant

SUMMARY:
In our country, although there is currently an emphasis on companion support within the scope of mother-friendly hospitals, there is no guide for companions. This study was planned to determine the effect of women who have companion support during labor on birth satisfaction, birth comfort, postpartum comfort level and positive birth outcomes, as well as the opinions of the people who provide support. Based on the results obtained and the positive contributions to maternal satisfaction during the labor process, birth and postpartum comfort process, mother-baby health, as well as the opinions of the companions, a 'Pregnant Support Guide in Labor' will be created and the companions will be enabled to support the pregnant woman in line with this guide. In addition, based on the opinions of the attendants, the researchers plan to develop the 'Birth Support Satisfaction Scale'.

DETAILED DESCRIPTION:
Type of research The study is a Randomized Controlled Mixed Method study. Research Design This study is a mixed method study planned to be conducted to evaluate the effect of companion support on the labor process and the opinions of companions, using a randomized controlled experimental design and in-depth individual interview method. This clinical trial will be registered at ClinicalTrials.gov. Reporting will be adhered to CONSORT for parallel group randomized studies. (CONSORT 2010, Access date: 10 August 2022). The research is planned to be carried out in the delivery room of Sakarya Training and Research Hospital between 01 March 2023 and 30 December 2024.

Where the Research Will Be Conducted The study will be carried out in the delivery room of Sakarya Training and Research Hospital. Pregnant women who have started labor are admitted to the delivery room by a doctor, and labor follow-up is carried out by midwives and assistant doctors under the supervision of a gynecologist. On average, around 350 vaginal births occur monthly. Since the hospital is not mother-friendly, a companion is not allowed to accompany the pregnant woman in routine practices.

Data Collection Stages The intervention and control groups will be informed about the research, and a personal information form will be applied to pregnant women and their companions who accept it.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women aged 37-42.
* Women who are planning to give birth vaginally during their first week of pregnancy.
* First-time pregnant women.
* Women with no vision, hearing, or communication problems.
* Women who can speak and express themselves in Turkish.
* Women who are willing to participate voluntarily in the study.

Exclusion Criteria:

* Pregnant women with multiple pregnancies.
* Women who are planned to give birth by cesarean section.
* Women with any complications during pregnancy.
* Women with chronic diseases.
* Pregnant women with verbal, mental, or other communication disabilities.
* Among the pregnant women included in the control or intervention group, those who:
* Received epidural analgesia.
* Experienced instrumental delivery (with vacuum or forceps).
* Had postnatal complications in the newborn.
* Had complications related to episiotomy (such as 3rd and 4th degree laceration, hematoma).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Birth Comfort Scale Score | At the time of cervical dilatation reaching 8 cm during the intrapartum period
  The Birth Comfort Scale is a tool designed to evaluate the level of comfort experienced by women during labor and delivery. The scale measures the influence of physical, psychological, and environmental factors on comfort during childbirth. It allows women to assess aspects such as physical ease, pain management, a sense of security, and environmental support during labor. Typically, the scale follows a 5-point Likert format, with each item scored from 1 to 5 (1: Strongly disagree, 5: Strongly agree). The total comfort score can range from a minimum of 10 to a maximum of 50.
  The scale demonstrates high internal consistency as measured by Cronbach's Alpha, with values typically ranging between 0.80 and 0.90, indicating that it is a reliable tool for assessing birth comfort.

SECONDARY OUTCOMES:
Postpartum Comfort Scale | Two hours postpartum
  The Postpartum Comfort Scale is designed to assess the comfort levels of women during the postpartum period. The scale evaluates comfort in three key areas: physical, psychological, and socio-cultural. It measures factors such as physical discomforts, emotional state, social support, and environmental influences during the postnatal period. The scale is typically structured as a 5-point Likert scale, with each item scored from 1 to 5 (1: Strongly disagree, 5: Strongly agree). The total score indicates whether the woman's postpartum comfort is low or high.
  The scale's Cronbach's Alpha is typically reported to be 0.85 or higher, indicating high reliability. This tool helps healthcare professionals better understand and address the needs of women during the postpartum period, leading to more effective interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Bihter Akın, Study Chair — Selcuk University
Locations (2):
- Turkey (Türkiye) (2):
  - Bihter Akın, Selçuklu, Konya
  - Selcuk University, Konya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Balcik Colak M, Akin B, Kalkan SC, Uslu Yuvaci H. Effects of labor support on pregnant women's childbirth comfort, satisfaction and postpartum comfort levels: a randomized controlled trial. BMC Pregnancy Childbirth. 2025 Jul 24;25(1):789. doi: 10.1186/s12884-025-07904-6. PMID 40707892